CLINICAL TRIAL: NCT05507268
Title: Predictive Nomogram for Postoperative Acute Kidney Injury in Older Patients Undergoing Noncardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-004
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Acute Kidney Injury
Keywords: prediction model; nomogram; older; noncardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- older patients undergoing noncardiac surgery: older patients (aged ≥65 years) scheduled for noncardiac surgery
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Postoperative acute kidney injury is associated increased risk of morbidity and mortality. Older patients are at high risk of developing postoperative acute kidney injury. However, the incidence and associations of postoperative acute kidney injury in older patients are not well understood. This study aims to develop and validate a predictive nomogram for postoperative acute kidney injury in older patients undergoing noncardiac surgery.

DETAILED DESCRIPTION:
Postoperative acute kidney injury (AKI) affects approximately 2% to 40% of patients undergoing cardiac and major noncardiac surgeries.

Older patients are more susceptible to renal impairment than younger patients. However, the incidence and associations of AKI in older patients are rarely understood.

Generally, in-depth knowledge of risk factors and thus able to identify patients at high risk to develop postoperative AKI is essential to optimize perioperative prevention and protection strategies.

In this retrospective study, the investigators intend to develop and validate a predictive model for postoperative using the identified risk factors.

The primary outcome is postoperative AKI, which according to the Kidney Disease: Improving Global Outcomes (KDIGO) criterion, is defined as an absolute increase in serum creatinine of 0.3 mg/dL within 48 hours or a 1.5-fold increase from preoperative baseline within 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older

Exclusion Criteria:

* Emergency operation
* Cardiac surgery
* Incomplete data
* Incomplete data
* Local anesthesia
* Preoperative renal failure or requirement for dialysis

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients (aged ≥ 65 years) undergoing noncardiac surgery from 2012-2019
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | 7 days after surgery
  an absolute increase in serum creatinine of 0.3 mg/dl within 48 hours or a 1.5-fold increase from preoperative baseline within 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Principal Investigator — The First Medical Center of Chinese PLA General Hospital
Locations (1):
- the First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided